CLINICAL TRIAL: NCT02716571
Title: Recruiting Blood Donor With Allogeneic Natural Killer Cell Which Will be Used for HCC After TACE
Brief Title: Recruiting Blood Donor With Allogeneic Natural Killer Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor,, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MG4101_HCC_Donor
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Subjects; Healthy Participants
MeSH Terms: interventions — Leukapheresis; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Donors (Other): Healthy Donors will given white blood cell and plasma
  Interventions: Other: Leukapheresis or Plasmapheresis

INTERVENTIONS:
Other: Leukapheresis or Plasmapheresis — Leukapheresis: Donate 5x10^9 white blood cells and 400 ml of plasma. Plasmapheresis: Donate 400ml of plasma.
  Donated white blood cell and plasma will be manufactured MG4101(allogeneic natural killer cell) to use for Hepatocellular carcinoma(HCC) patients after Transarterial Chemoembolization(TACE).

SUMMARY:
This study on manufacture of MG4101 (allogeneic natural killer cell) to use for Hepatocellular carcinoma(HCC) after Transarterial Chemoembolization(TACE) will be harvested WBC(white blood cell) and plasma from healthy donors, or plasma from healthy donors by leukapheresis or plasmapheresis procedure.

DETAILED DESCRIPTION:
The purpose of this study is to manufacture MG4101 (allogeneic natural killer cell) which will be used for clinical trial in HCC after TACE.

Manufacturing MG4101 involves WBC(white blood cell) and plasma harvesting from healthy donors. Another methodology for plasma harvesting can be performed through the leukapheresis procedure.

Healthy donors were requested to visit the institution twice for receiving either leukapheresis or plasmapheresis procedure. During the screening, study participants (subjects) were given a written informed consent, which was written in accordance with the Declaration of Helsinki and regional laws. Following the screening, study participants (subjects) each received a questionnaire for medical examination and a preliminary examination to evaluate their suitability as donors.

If the study subjects' test result is suitable for clinical study standards either leukapheresis or plateletpheresis process will be performed for the following three weeks.

The MG4101 will be manufactured from harvesting WBC and plasma, under the conditions of both GMP(Good Manufacturing Practice) at Green Cross Lab Cell Corp. (Korea). Also, the resulting MG4101, will be cryopreserved for using clinical trial in HCC after TACE.

ELIGIBILITY:
Inclusion Criteria:

* Male body weight must be over 50 ㎏, Female body weight must be over 45㎏,
* Temperature less than 37.5 Celsius,
* Systolic blood pressure greater than 90 and less than 180 ㎜Hg,
* Diastolic blood pressure less than 100 ㎜Hg,
* Heart rate between 50 to 100 beats per minute.
* No abnormality in CBC(complete blood count) and PT/aPTT(prothrombin time /activated Partial Thromboplastin Time)Test
* ALT(ALanine Transaminase) Less than 65IU/L
* No history of bleeding and bleeding diathesis

Exclusion Criteria:

* Drinking more than 3 alcoholic drinks per week.
* Under the 12.5g/dl hemoglobin (38% packed cell volume)
* Positive tests for blood borne pathogens (HBV, HCV(Hepatitis C Virus), HIV, HTLV(human T lymphotropic virus)-I,II, syphilis, CMV(Cyto-Megalo-Virus), EBV(Epstein-Barr Virus))
* Person who falls short of health standards, such as a patient with an infectious disease or a patient who take medication, who is prescribed by Ordinance of the Ministry of Health and Welfare as unfit to donate blood.
* Donor taking prescription medications other than those deemed allowable by the investigator.

  * Aspirin within prior 3 days
  * Ticlopidine within prior 2 weeks
  * Isotretinoin, Finasteride within prior 1 month
  * Dutasteride within prior 6 months
* Hepatitis B immune globulin(HBIG), Placental Extract within prior 1 year
* People vaccinate against Cholera, diphtheria, influenza, A hepatitis, B hepatitis, typhoid, poliomyelitis, Japanese encephalitis, tetanus, pertussis, Korean hemorrhagic fever, Bacillus anthracis, rabies virus cannot donate blood for 24 hours.
* People vaccinate against measles, epidemic parotitis, yellow fever and administer Oral Polio-Vaccine, Oral Poliomyelitis Vaccine cannot donate blood for 2 weeks.
* People vaccinate against rubella virus, varicella virus, BCG cannot donate blood for 1 month.
* If female, pregnant or parturition or miscarriage within prior 6 months
* Transfusion within prior 1 years
* A Whole blood donation within prior 2 months.
* A Plasmapheresis, a plateletpheresis and a 2 units plateletpheresis within the prior 14 days
* A Leukapheresis within prior 72 hours
* Having received more than 5 whole blood donation within prior 1 years

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Ex vivo expended Allogeneic Natural killer cells(MG4101) viability | 21 days
Purity of ex vivo expended Allogeneic Natural killer cells(MG4101) | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Lim O, Lee Y, Chung H, Her JH, Kang SM, Jung MY, Min B, Shin H, Kim TM, Heo DS, Hwang YK, Shin EC. GMP-compliant, large-scale expanded allogeneic natural killer cells have potent cytolytic activity against cancer cells in vitro and in vivo. PLoS One. 2013;8(1):e53611. doi: 10.1371/journal.pone.0053611. Epub 2013 Jan 11. PMID 23326467